CLINICAL TRIAL: NCT04309097
Title: Reducing Eye Strain and Anxiety Using a Digital Intervention During Online Learning Class Recess Among Children at Home: A Randomized Controlled Trial
Acronym: RESILIENT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Sun Yat-sen University (Other)
Responsible Party: Principal Investigator, Yingfeng Zheng, Professor, Sun Yat-sen University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2020KYPJ045
Record Dates: First submitted 2020-03-11; First posted 2020-03-16 (Actual); Last update posted 2020-05-12 (Actual); Status verified 2020-05

CONDITIONS: Anxiety; Digital Eye Strain
MeSH Terms: conditions — Anxiety Disorders

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Digital intervention (Experimental): Participants will have access to a live-streaming App that offers Recess and Exercise Advocate Program (REAP).
  Interventions: Behavioral: Digital intervention
- Information-only intervention (Active Comparator): Participants will have access to health information only.
  Interventions: Behavioral: Information-only intervention

INTERVENTIONS:
Behavioral: Digital intervention — REAP is a live-streaming platform that allows users to shoot short videos or photos related to their physical exercise or eye relaxation (e.g., staring out of the window) using their smartphones. The app has been optimised to be used with the iPhone or Android.
  When taking a online course recess, students will have access to the REAP platform that allows them to watch stay-at-home workout videos developed by exercise physiologists. Students will then be asked to create their own workout videos/photos and upload them to the live-streaming platform. When upload is completed, students will receive instant motivational messages to increase their engagement with the program.
  Arms: Digital intervention
Behavioral: Information-only intervention — Participants will have access to online health information and stay-at-home workout videos.
  Arms: Information-only intervention

SUMMARY:
The primary aim of the current study is to conduct a cluster-randomized control trial to evaluate the effectiveness of a novel digital intervention in reducing anxiety and digital eye strain compared to usual care among Chinese children during the period of home confinement.

DETAILED DESCRIPTION:
In response to the coronavirus disease 2019 (COVID-19), many countries have taken the decision of school closure after the confirmation of coronavirus cases in the general population. In China, the burden of COVID-19 is among the highest in the world, with more than 80,000 cases confirmed by 11th March 2020. An estimate of 220 million children and adolescents are confined at home for weeks with inadequate level of physical activity and more susceptible to anxiety. There is also a concern of digital eye strain for many children who spend hours daily in front of a computer screen for recreation or learning purposes.

Recess represents an essential scheduled period in a school day for psychological and physical relaxation. During the unusual period of home confinement, many schools have already issued physical activity requirement and policy recommending recess and physical activity breaks. However, recess could be easily skipped by students during online learning at home.

Mobile health intervention offers a potential opportunity for capitalizing on digital technology as a feasible modality to encourage recess activities, especially in regions where social distancing is implemented as an emergency measure. The primary aim of the current study is to conduct a cluster-randomized control trial to evaluate the effectiveness of a novel digital intervention during recess in reducing anxiety and digital eye strain compared to usual care among Chinese children during the period of home confinement.

ELIGIBILITY:
Inclusion Criteria:

* Grade 7 (12-13 years old) students in Duanzhou District, Zhaoqing city
* Students under home confinement and enrolled in online learning courses, during the COVID-19 outbreak

Exclusion Criteria:

* Autism Spectrum Disorders and Pervasive Developmental Delay or Disorder
* Mental Retardation
* Psychotic Disorders and Schizophrenia
* Mania or Hypomania disorders
* Suicidal behavior and/or acute plan that require higher level of care
* Participation in psychotherapy

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 954 (Actual)
Dates: Start 2020-03-16 (Actual); Primary Completion 2020-03-29 (Actual); Study Completion 2020-03-29 (Actual)

PRIMARY OUTCOMES:
Change in anxiety | Baseline & at 2 weeks
  Change in anxiety will be measured by the Spence Children's Anxiety Scale (SCAS) designed by Spence (1998). The SCAS (45-item) is self-report scale with a 4-point Likert type, consisting of 44 items and one open-ended question. Overall assessment is done by total score.

SECONDARY OUTCOMES:
Change in syndromes of digital eye strain | Baseline & at 2 weeks
  Syndromes of digital eye strain will be measured with the Computer Vision Syndrome Questionnaire (CVS-Q) designed by Seguí et al (2015). The self-reported CVS-Q questionnaire (16-item) evaluates the frequency (never, occasionally or often/always) and the intensity (moderate or intense) of 16 symptoms: burning, itching, feeling of a foreign body, tearing, excessive blinking, eye redness, eye pain, heavy eyelids, dryness, blurred vision, double vision, difficulty focusing for near vision, increased sensitivity to light, colored halos around objects, feeling that sight is worsening, and headache. Overall assessment is done by total score.
Change in sleeping quality | Baseline & at 2 weeks
  The PROMIS pediatric sleep disturbance questionnaire (4-item), designed by Forrest et al (2018), assesses self-reported experiences of sleep disturbance over the past 7 days. Raw score will be converted to T-Score.
Changes in time (hour) spent on different near work activities | Baseline & at 2 weeks
  Participants will be asked to indicate the average time in hours per day spent on each the following activities: reading, writing, computer/PAD use, smart phone, watching TV, and playing video games.

CONTACTS AND LOCATIONS:
Locations (1):
- Secondary schools, Zhaoqing, Guangdong, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Wang G, Zhang Y, Zhao J, Zhang J, Jiang F. Mitigate the effects of home confinement on children during the COVID-19 outbreak. Lancet. 2020 Mar 21;395(10228):945-947. doi: 10.1016/S0140-6736(20)30547-X. Epub 2020 Mar 4. No abstract available. PMID 32145186
- [Background] Segui Mdel M, Cabrero-Garcia J, Crespo A, Verdu J, Ronda E. A reliable and valid questionnaire was developed to measure computer vision syndrome at the workplace. J Clin Epidemiol. 2015 Jun;68(6):662-73. doi: 10.1016/j.jclinepi.2015.01.015. Epub 2015 Jan 28. PMID 25744132
- [Background] Forrest CB, Meltzer LJ, Marcus CL, de la Motte A, Kratchman A, Buysse DJ, Pilkonis PA, Becker BD, Bevans KB. Development and validation of the PROMIS Pediatric Sleep Disturbance and Sleep-Related Impairment item banks. Sleep. 2018 Jun 1;41(6). doi: 10.1093/sleep/zsy054. PMID 29546286
- [Background] Spence SH. A measure of anxiety symptoms among children. Behav Res Ther. 1998 May;36(5):545-66. doi: 10.1016/s0005-7967(98)00034-5. PMID 9648330
- [Derived] Zheng Y, Wang W, Zhong Y, Wu F, Zhu Z, Tham YC, Lamoureux E, Xiao L, Zhu E, Liu H, Jin L, Liang L, Luo L, He M, Morgan I, Congdon N, Liu Y. A Peer-to-Peer Live-Streaming Intervention for Children During COVID-19 Homeschooling to Promote Physical Activity and Reduce Anxiety and Eye Strain: Cluster Randomized Controlled Trial. J Med Internet Res. 2021 Apr 30;23(4):e24316. doi: 10.2196/24316. PMID 33882021